CLINICAL TRIAL: NCT02976415
Title: CardiO Cycle: A Pilot Safety and Feasibility Study of In-Bed Cycling in Patients Post Cardiac Surgery
Brief Title: In-Bed Cycling in ICU Patients Post Cardiac Surgery
Acronym: CardiO Cycle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Anastasia Newman, Physiotherapist, PhD Student, Hamilton Health Sciences Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-1999-GRA
Record Dates: First submitted 2016-11-08; First posted 2016-11-29 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Cardiac Disease; Critical Illness; Critical Illness Polyneuropathy; Critical Illness Myopathy; Thoracic Surgery
Keywords: Cardiac Surgery; Physiotherapy; In-Bed Cycling; Mechanical Ventilation; Cycle Ergometry; Early Mobilization; Rehabilitation; Critical Care; Intensive Care Unit
MeSH Terms: conditions — Heart Diseases; Critical Illness; Polyneuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: In-Bed Cycling — 20 minutes of in-bed cycling, either active, passive or a combination of active and passive.
  Other Names: Bedside Cycling; Bedside Ergometry

SUMMARY:
The purpose of this study is to determine if in-bed cycling is safe and feasible in critically-ill patients after open heart surgery. The investigators hypothesize that in-bed cycling can be safely used with this population and that it is feasible to use in a fast-paced cardiac intensive care unit.

DETAILED DESCRIPTION:
Background: Advances in medical science and technologies have lead to more effective management of critically-ill patients with a subsequent improvement in ICU survival rates. Patients who survive their ICU stay are often left with post-ICU impairments including muscle weakness and functional limitations. Cardiac surgeries are commonly performed worldwide with the majority of patients requiring post-operative ICU care. In the past decade, patients who qualify for cardiac surgery tend to be older, have a great number of co-morbidities and are more likely to require a prolonged ICU stay. The effectiveness of physiotherapy and various rehabilitation modalities in patients both pre- and post cardiac surgery has been investigated. However, to date no study specifically addresses the feasibility and safety of in-bed cycling in patients undergoing cardiac surgery who require prolonged critical care.

Principle Research Question: Is in-bed cycling a safe and feasible intervention in patients post cardiac surgery that require a prolonged stay in critical care?

Methods: Adult patients post-cardiac surgery admitted to the cardiac surgery ICU who will remain intubated and ventilated for at least 72 hours will be eligible for enrollment. Participants will receive 20 minutes of in-bed cycling plus routine physiotherapy performed by critical care physiotherapists. Patients will be enrolled for 28 days or until they are able to ambulate.

Primary Outcomes: Safety of bedside cycling will be evaluated by monitoring the number of adverse events that occur during each cycling session. Feasibility of implementing in-bed cycling into daily physiotherapy practice will be evaluated by determining if cycling sessions can be conducted at least eighty percent of the time that cycling is appropriate.

Relevance: Before conducting a larger randomized controlled trial investigating the effectiveness of in-bed cycling in the critically-ill cardiac surgery population, the safety of this intervention needs to be determined. This will be the first study in a program of research evaluating bedside cycling in the cardiac surgical ICU.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults patients aged 18 years and greater
* History of cardiac surgery in the past seven days
* Admitted to the cardiac surgery ICU for greater than 3 days but less than 7 days
* Mechanically ventilated for at least 72 hours and expected to remain ventilated for at least two more days
* Able to ambulate independently, with or without a gait aid, prior to hospital admission

Exclusion Criteria:

* Uncomplicated post-operative course with expected discharge to ward within 24 to 72 hours
* Previous lower extremity amputation
* Open or unstable saphenous vein graft sites
* Inability to understand English
* Body size and/or weight that is incompatible with the bedside ergometer
* Patients who are not expected to survive their ICU stay

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Number of safety events that occur during cycling sessions | From date of study enrollment until the date of study completion, up to 28 days maximum
  Potential safety events include:
  * Hypertension (systolic blood pressure greater than 160 mmHg)
  * Hypotension (systolic blood pressure less than 90 mmHg)
  * Oxygen desaturation to less than 85% for more than two minutes
  * Cardiorespiratory arrest
  * Removal of any lines or tubes (chest tubes, pulmonary artery catheter, nasal-gastric tube, Jackson-Pratt drains, central venous catheter, endotracheal tube, tracheostomy decannulation)
  * New onset cardiac arrhythmias (atrial fibrillation, bigeminy, trigeminy, junctional, heart block rhythms)
  * Saphenous vein graft dehiscence
  * New onset agitation
Feasibility of completing 80% of eligible cycling sessions | From date of study enrollment to the date of study completion, up to 28 days maximum
  The feasibility of implementing in-bed cycling into daily physiotherapy practice will be evaluated by determining if cycling sessions can be conducted at least 80% of the time that cycling is appropriate.

SECONDARY OUTCOMES:
Feasibility of Completing Hand Grip Strength at ICU Awakening and ICU Discharge | When patient awake (unspecified time, patient dependent), at completion of study involvement (maximum: day 28 of ICU)
  Hand grip strength will be assessed using a hand-held JAMAR dynamometer. Patients will be seated with elbow bent to 90 degrees. Patients will be asked to "squeeze the handle as hard as possible" and the maximum score will be taken after five seconds. Average of three trials will be documented.
Two Minute Walk Test | At ICU Awakening (an estimated 8 days after study enrollment) and at the completion of the study (maximum: day 28 of ICU)
  In an unobstructed area, patients will be instructed to walk back and forth covering as much distance as possible in two minutes. Gait aids may be used and patients are permitted to rest as needed during the test. No encouragement will be provided during the two minute test. The number of rest stops, the duration of the rests and the distance traveled in meters will be documented.
Functional Status Score for the ICU (FSS-ICU) | Assessed daily, up to a maximum of 28 days
  The FSS-ICU is a five-item functional measure that evaluates the ability of each client to perform five specific tasks (rolling, supine to sit, sitting at edge of bed, sit to stand, walking). Each scale is assessed using an 8-point ordinal scale (0 - inability to perform the task to 7 - able to perform the task independently)

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia N Newman, PhD Student, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton General Hosptial, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Newman ANL, Kho ME, Harris JE, Zamir N, McDonald E, Fox-Robichaud A, Solomon P; Canadian Critical Care Trials Group. CardiO Cycle: a pilot feasibility study of in-bed cycling in critically ill patients post cardiac surgery. Pilot Feasibility Stud. 2021 Jan 7;7(1):13. doi: 10.1186/s40814-020-00760-5. PMID 33407923